CLINICAL TRIAL: NCT04625257
Title: COVID-19 in Baselland: Validation of Simple and Accurate Tests for COVID-19 Detection, Monitoring and Tracing (ACCURATE-BL-COVID-19)
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: ETH Zurich Department for Biosystems, Science and Engineering (Unknown); Kanton Basel- Landschaft (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-01112; ch20Savic2
Record Dates: First submitted 2020-11-10; First posted 2020-11-12 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Coronavirus Infectious Disease 2019 (COVID-19)
Keywords: severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2); quantitative reverse transcription polymerase chain reaction (qRT-PCR) assay; point of care tests (POCT); next-generation sequencing (NGS) method; contact tracing; transmission chains; crude RNA extraction from saliva; loop mediated amplification (LAMP) assay; viral nucleic acid analysis platform
MeSH Terms: conditions — COVID-19 | interventions — Antibody Formation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biological material is appropriately stored in a restricted area only accessible to authorized personnel. Until completion of the study, the material will be stored in the biobank "SERO-BL-COVID-19".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Saliva based assay: crude RNA extraction — Crude RNA extraction to inactivate the virus and stabilize the RNA for transport at room temperature. Validation of the crude RNA extraction from saliva in combination with NGS diagnostics and LAMP assays and point of care test (POCT) for rapid detection of viral antigens on patients' samples.
Other: Validation of the NGS method — Compare the results obtained with the next-generation sequencing (NGS) method to the nasopharyngeal swabs analysed in a FAMH certified lab.
Other: Validation of the LAMP assays — The RNA will be analyzed onsite using the loop mediated amplification (LAMP) assay.
Other: Validation of the POCT Antigen and Antibody tests — Rapid point of care tests (POCT) detecting viral protein antigens (Ag) and antibodies (Ab) on patients' samples. POCT are often employed in low income countries, but for COVID-19 they are not yet characterized. Their performance is to be characterized that they can be used as a safe guard if the lab diagnostics fail.

SUMMARY:
This study is to establish an accurate, robust and easily scalable COVID-19 viral nucleic acid analysis platform from, but not limited to, saliva to help enable and support contact tracing in the canton of Baselland/ Switzerland. To achieve this, crude ribonucleotide acid (RNA) extraction from saliva is validated in combination with next-generation sequencing (NGS) diagnostics and loop mediated amplification (LAMP) assays as well as point of care test (POCT) for rapid detection of viral antigens on patients' samples.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic patients getting tested for COVID-19

Exclusion Criteria:

* mentally incompetent adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic patients arriving at the COVID-19 test center Feldreben in Muttenz, Basel Land and at Swiss TPH in Basel, Basel Stadt to get tested for COVID-19.
Sampling Method: Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2020-10-24 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
qualitative method validation of the crude extraction in combination with the LAMP or the NGS (count values for detection) | single point assessment at baseline
  For all qualitative method validation, the qualitative and quantitative result of the Foederatio Analyticorum Medicinalium Helveticorum (FAMH) performed RT-PCR (patient does / does not have SARS-Cov-2 and if yes, how many "ct" values for detection) is considered as the gold standard against which the crude extraction in combination with the LAMP or the NGS method using univariate measures is compared.

CONTACTS AND LOCATIONS:
Overall Officials: Miodrag Savic, Dr. med. Dr. med. dent., Principal Investigator — Cantonal Office of Public Health, Economics and Health Directorate, Canton Basel-Landschaft
Locations (1):
- Cantonal Office of Public Health, Economics and Health Directorate, Canton Basel-Landschaft, Liestal, Switzerland